CLINICAL TRIAL: NCT01429870
Title: A Phase IV, Randomized, Double Blind, Placebo Controlled, Single-center Study of the Impact of Topical Steroids on Narrow Band UVB (Ultraviolet B) and Dithranol Combination Treatment of Psoriasis (DIPSO)
Brief Title: Steroids Added to Dithranol and Narrow Band UVB(Ultraviolet B) (UVBnb) in Psoriasis
Acronym: DIPSO
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DIPSO; KEK-ZH 2010-0171-5 (Other: Ethical committee Zurich)
Record Dates: First submitted 2011-08-18; First posted 2011-09-07 (Estimated); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Triamcinolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Steroid active treatment (Active Comparator): Triamcinolone acetonide 0.1% in unguentum leniens topically
  Interventions: Drug: Steroid active treatment
- Vehicle (Placebo Comparator): unguentum leniens topically
  Interventions: Drug: Steroid active treatment

INTERVENTIONS:
Drug: Steroid active treatment — Triamcinolone in unguentum leniens 0.1%
  Other Names: Topical triamcinolone

SUMMARY:
Objective(s):

(i) To assess the effect of adjunctive topical steroids in the combined treatment with UVBnb and dithranol on the remission time after therapy till a relapse of psoriasis defined as 50% loss of PASI (Psoriasis Area and Severity Index) improvement obtained through the antecedent treatment.

(ii) To assess the impact of adjuvant topical steroids in the combined treatment with UVBnb and dithranol on the clearing time of psoriasis lesions under therapy (PASI 75).

* Trial with medicinal product

DETAILED DESCRIPTION:
(i) To assess the effect of adjunctive topical steroids in the combined treatment with UVBnb and dithranol on the remission time after therapy till a relapse of psoriasis defined as 50% loss of PASI (Psoriasis Area and Severity Index) improvement obtained through the antecedent treatment.

(ii) To assess the impact of adjuvant topical steroids in the combined treatment with UVBnb and dithranol on the clearing time of psoriasis lesions under therapy (PASI 75).

* Trial with medicinal product

ELIGIBILITY:
Inclusion criteria:

* Moderate to severe psoriasis of the chronic-plaque and / or guttata type

Exclusion criteria:

* Participation in a Goeckerman therapy regimen within 6 months previous to the present study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Relapse 50% PASI after treatment, time to PASI 75% on treatment | 2 years
  Relapse 50% PASI after treatment, time to PASI 75% on treatment

CONTACTS AND LOCATIONS:
Overall Officials: Guenther Hofbauer, MD, Principal Investigator — University Hospital Zurich, Division of Dermatology
Locations (1):
- University Hospital Dermatology Department, Zurich, Switzerland